CLINICAL TRIAL: NCT03229044
Title: Tetranectin as a Novel Obesity-associated Adipokine for Regulating Lipid Accumulation
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 9461701203
Record Dates: First submitted 2017-07-13; First posted 2017-07-25 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2005-12

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: adipokine, tetranectin, lipid metabolism, body mass index
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — tetranectin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Adipose tissues from breast were preserve in -80 refrigerator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- BMI 18-21: Tetranectin mRNA and protein level were measure in the adipose tissues which were belonging to body mass index is 18-21 kg/m2
  Interventions: Genetic: Tetranectin
- BMI 33-39: Tetranectin mRNA and protein level were measure in the adipose tissues which were belonging to body mass index is 33-39 kg/m2
  Interventions: Genetic: Tetranectin
- BMI 25-30: Tetranectin mRNA and protein level were measure in the adipose tissues which were belonging to body mass index is 25-30 kg/m2
  Interventions: Genetic: Tetranectin

INTERVENTIONS:
Genetic: Tetranectin — Adipose tissues were obtained from the breast of breast cancer patients with 0 to 1 progression stage. The subjects were 33-51 y of age (mean = 43.6, SD = 6.2) with a BMI of 16-33 kg/m2 (mean = 21.5, SD = 4.5). Blood samples were collected after an overnight fasting. Serum was separated by centrifugation and stored at -80 ℃ until analysis. Plasma Tetranectin,triglyceride (TG), high density lipoprotein (HDL), low density lipoprotein (LDL), cholesterol, glucose and insulin were measured. And the tetranectin mRNA and protein level was measure in adipose tissue

SUMMARY:
Adipose tissue is strongly correlated to obesity and diabetes which are two major problems in the worldwide. Adipose tissue is involved in modulating glucose and energy metabolism locally and systemically by secreting factors, called adipocytokines. Tetranectin (TN), a novel adipocytokine, is secreted by adipose tissues. TN may regulate the glucose/energy homeostasis to affect lipid accumulation.The role of TN in adipocytes with or without TN on regulation of adipose tissue growth and lipid metabolism is valuable to be studied.

Materials and methods: Secreted proteins from human adipocyte culture medium were deciphered using 2-D polyacrylamide gel electrophoresis and determined by LC/MS with MALDI-TOF analysis of proteins. Adipose tissues were obtained from the breast of 15 women undergoing mastectomy. Serum samples from 200 normal healthy people and 54 breast cancer patients were assigned to either a lean or obese group according to the body mass index. The TN protein concentration was measured in the culture medium of stromal-vascular fraction (SVF)-derived adipocytes from healthy humans, breast cancer patients, pigs and also from 3T3-L1 cells. Associations between plasma TN and other biomarkers were assessed with Pearson's correlations and multivariable linear regression.

DETAILED DESCRIPTION:
Adipose tissues were obtained from the breast of breast cancer patients with 0 to 1 progression stage. All participants gave permission and the study was approved by the Ethics Committee of National Taiwan University Hospital as no. 9461701203.

From 2012 to 2013 in National Taiwan University Hospital, a cross-sectional sampling of 21 to 78 -year old people included women and men who were living in Taiwan. Blood samples were collected after an overnight fasting. Serum was separated by centrifugation and stored at -80 ℃ until analysis. Plasma triglyceride (TG), high density lipoprotein (HDL), low density lipoprotein (LDL), cholesterol, glucose and insulin were measured. Fasting serum samples were obtained from 193 randomly selected persons having health check-ups. To investigate the relationship among TN and breast cancer, fasting serum samples also obtained from 54 randomly selected breast cancer patients who were 25 to 59 years old with elected surgery for breast cancer stage 0 and 1.

ELIGIBILITY:
Inclusion Criteria:

1. Must be above age 20 years old.
2. Subjects must sign the written informed consent form.
3. Must have residual fat after surgery.
4. Clinical diagnosis of liposuction and tumor resection.

Exclusion Criteria:

1. Terminal cancer.
2. Subjects have no fat tissue after surgery.
3. Pregnant subjects.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adipose tissues were obtained from the breast of breast cancer patients with 0 to 1 progression stage.
Sampling Method: Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2005-12-06 (Actual); Primary Completion 2008-12-05 (Actual); Study Completion 2008-12-05 (Actual)

PRIMARY OUTCOMES:
Tetranectin expression measure | through study completion, an average of 2 years
  Detect Tetranectin expression in adipose tissue by qPCR or Western blotting

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Torng Ding, Ph D, Principal Investigator — National Taiwan University

IPD SHARING:
Plan to Share IPD: Undecided
Serum samples and adipose tissue from breast cancer patients were assigned to either a lean or obese group according to the body mass index. The TN protein concentration was measured in the serum samples and culture medium of stromal-vascular fraction (SVF)-derived adipocytes from breast cancer patients,

REFERENCES:
- [Background] Jaquinod M, Holtet TL, Etzerodt M, Clemmensen I, Thogersen HC, Roepstorff P. Mass spectrometric characterisation of post-translational modification and genetic variation in human tetranectin. Biol Chem. 1999 Nov;380(11):1307-14. doi: 10.1515/BC.1999.166. PMID 10614823
- [Background] Iba K, Durkin ME, Johnsen L, Hunziker E, Damgaard-Pedersen K, Zhang H, Engvall E, Albrechtsen R, Wewer UM. Mice with a targeted deletion of the tetranectin gene exhibit a spinal deformity. Mol Cell Biol. 2001 Nov;21(22):7817-25. doi: 10.1128/MCB.21.22.7817-7825.2001. PMID 11604516